CLINICAL TRIAL: NCT03174990
Title: The Effect of Aspirin and Thienopyridine Non-responsiveness on Outcomes in Peripheral Arterial Disease
Brief Title: Aspirin and Thienopyridine Resistance in Peripheral Arterial Disease
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Khung Keong Yeo, MD, Staff physician, University of California, Davis
Other Study IDs: 224399
Record Dates: First submitted 2017-05-25; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Peripheral Arterial Disease; Clopidogrel, Poor Metabolism of
Keywords: aspirin; clopidogrel; peripheral arterial disease; genetics
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Aspirin responsive: The participant is shown to be responsive to platelet activity inhibition by aspirin, as determined by testing with VerifyNow
- Aspirin non-responsive: The participant is shown to be non-responsive to platelet activity inhibition by aspirin, as determined by testing with VerifyNow
- Clopidogrel responsive: The participant is shown to be responsive to platelet activity inhibition by clopidogrel, as determined by testing with VerifyNow
- Clopidogrel non-responsive: The participant is shown to be responsive to platelet activity inhibition by clopidogrel, as determined by testing with VerifyNow

SUMMARY:
This study evaluates the effects of Aspirin and thienopyridine resistance in relation to clinical cardiovascular outcomes as the genetic predictors of, and outcomes associated with aspirin and thienopyridine resistance in patients with peripheral arterial disease (PAD) currently remain unknown.

DETAILED DESCRIPTION:
Although anti-platelet therapy is a cornerstone of PAD treatment, the investigators know very little about the prevalence, genetic determinants and clinical relevance of aspirin and thienopyridine resistance in PAD patients. The investigators expect to report on the prevalence of, and impact on outcomes from aspirin and/or thienopyridine (eg. clopidogrel) resistance, in patients who undergo peripheral arterial angiography/interventions (including carotid angiography/interventions) and operations. This study will provide important information on the utility of testing for aspirin and thienopyridine resistance and improve understanding of the genetic and pathophysiologic basis of anti-platelet therapy resistance in patients with cardiovascular disease, including PAD. Most importantly, this study will serve as the basis for a subsequent randomized prospective trial of different treatment options in PAD patients with aspirin/thienopyridine resistance.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing PAD (carotid or lower extremity) angiography or intervention
* greater than or equal to 18 years of age

Exclusion Criteria:

* patient unable to take aspirin and thienopyridine for any reason (not excluded if take at least one of either medication)
* hematocrit less than or equal to 30%
* hematocrit greater than or equal to 52%

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients enrolled between August 2010 and September 2012, with angiographically documented PAD involving carotid or lower extremity arteries. Patients may have been treated surgically or endovascularly at the discretion of the primary physician.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2010-08-31 (Actual); Primary Completion 2013-05-17 (Actual); Study Completion 2013-12-20 (Actual)

PRIMARY OUTCOMES:
Clopidogrel non-responsiveness | Immediate
  Clopidogrel non-responsiveness was defined as patients with Plavix reaction units (PRU) ≥ 235
Aspirin non-responsiveness | Immediate
  Aspirin non-responsiveness was defined as patients with aspirin reaction units (ARU) ≥ 550
Composite of major adverse cardiovascular events | 1 year
  Composite of major adverse cardiovascular events including all-cause mortality, myocardial infarction, stroke, target vessel revascularization (TVR) and limb loss in patients who underwent extremity intervention.

SECONDARY OUTCOMES:
Genetic predictors of aspirin and clopidogrel non-responsiveness | Immediate
  Single nucleotide polymorphisms (SNP) were correlated to measures of aspirin and clopidogrel non-responsiveness

CONTACTS AND LOCATIONS:
Overall Officials: khung keong, MD, Principal Investigator — Cardiovascular interventionalist
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No